CLINICAL TRIAL: NCT02857244
Title: A Multidisciplinary Approach to Manage Gait Difficulty in Parkinson Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Site did not obtain LIRB approval due to medication usage.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1577
Record Dates: First submitted 2016-07-25; First posted 2016-08-05 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease
Keywords: Freezing of Gait
MeSH Terms: conditions — Parkinson Disease | interventions — Duloxetine Hydrochloride; Donepezil; Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Treatment Arm (Other): Each patient will take Duloxetine 30mg for 1 week, followed by 60mg qam for 1 week, 90mg qam for 1 week, and 120mg qam for 1 week, if tolerated. The patient will be taking Duloxetine for a total of 4 weeks. The dose of Duloxetine will be reduced if the patient cannot tolerate. Donepezil will then be added to Duloxetine 120mg qam (or the highest dose the patient can tolerate) by 5mg qd for 1 week, followed by 10mg qd for 1 week.
  After a 4-week washout period, each patient will take Modafinil 100mg qam for one week, followed by 200mg qam for 1 week.
  Patients will come into the medical center on 5 occasions, 1 for screening/baseline, 1 after completion of duloxetine, 1 after completion of duloxetine+donepezil, 1 after four-week washout, 1 after completion of modafinil.
  Interventions: Drug: Duloxetine; Drug: Donepezil; Drug: Modafinil

INTERVENTIONS:
Drug: Duloxetine — Patients will first receive Duloxetine for 4 weeks starting at 30mg, 60mg, 90mg then 120mg (if tolerated). Increases in dosage amounts will occur every week.
Drug: Donepezil — Patients will receive Donepezil after 4 weeks of dosing with Duloxetine. Patients will receive Donepezil in combination with the highest dose of Duloxetine that was tolerated. Patients will remain on this for 2 weeks with increasing doses at each week. One week of 5mg, one week of 10mg.
  Other Names: Aricept
Drug: Modafinil — Patients will receive Modafinil after a 4 week washout period (after dosing with donepezil & duloxetine in combination). Patients will receive Modafinil for two weeks with increasing doses at each week. One week at 100mg, one week at 200mg.

SUMMARY:
The study team proposes to treat Parkinson's patients with gait difficulty with multidisciplinary approach of medications. Single medication treatment, such as the use of cholinergic-boosting anti-dementia medication targeting cholinergic deficiency to improve executive dysfunction and attention deficit, or the use of medication boosting the norepinephrine system, have not proven effective so far in treating the gait difficulty. Anti-anxiety medications, particularly the SNRI (serotonin and norepinephrine reuptake inhibitor) medications, which also ameliorate the norepinephrinergic deficiency, have not been studied except for one successful case report using duloxetine to treat primary progressive freezing of gait.

Targeting multiple mechanisms at same time, such as the combination of a SNRI antianxiety medication (also boosting the norepinephrine system, such as duloxetine) with an anti-dementia medication correcting the cholinergic deficiency (such as donepezil), or targeting a new mechanism, such as the use of anti-GABAergic medication targeting the area responsible for gait and sleep cycle (pedunculopontine nucleus area, PPNa) should be tried.

Therefore, a collaboration of multidisciplinary teams among the neurology movement disorder team and cognition and sleep team, and psychiatry team is essential, which has not been tried before in studying and treating the challenging gait difficulty in Parkinson patients.

DETAILED DESCRIPTION:
The study team proposes to treat parkinsonian patients with gait difficulty of FOG with the SNRI anti-anxiety medication duloxetine for 4 weeks, followed by an additional anti-dementia medication donepezil for 2 weeks to determine whether antianxiety treatment alone or in combination with the anti-dementia medication can improve gait. Another medication with GABA antagonist property targeting the gait controlling area PPNa (and improving anxiety and cognition as well), modafinil, will be tried for 2 weeks after a 4-week washout period of the previous medications.

Specifically, the investigators will propose an open label prospective pilot study using duloxetine to treat 22 parkinsonian patients with FOG, aiming for estimated 80% power of detecting 50%. Each patient will take duloxetine 30mg for 1 week, followed by 60mg qam for 1 week, 90mg qam for 1 week, and 120mg qam for 1 week, if tolerated. The patient will be taking duloxetine for a total of 4 weeks, as described above. The dose of duloxetine will be reduced if the patient cannot tolerate a higher rank dose as designated. This principle will apply to the other two medications used in the study as well. Donepezil will then be added to duloxetine 120mg qam (or the highest dose the patient can tolerate if it is lower than 120mg) by 5mg qd for 1 week, followed by 10mg qd for 1 week. Each patient will visit us 3 times (baseline and at the end of each medication, namely 4 weeks after the duloxetine and 2 weeks after the donepezil), checking UPDRS-III (and PSP scale as well for PSP patients), stand-walk-sit, freezing of gait questionnaire, Montreal cognitive scale (MoCA) for patients before and after Donepezil treatment, and anxiety scale for patients before and after duloxetine treatment (if the patient is on dopaminergic medication). Daily falls, freezing of gait (by the questionnaire) and quality of life (by PDQ-39 scale) over the past week prior to the clinical visit will also be checked.

After a 4-week washout period, each patient will take modafinil 100mg qam for 1 week, followed by 200mg qam for 1 week. Each patient will visit us twice (baseline at the end of the 4-week washout period, and at the end of the 2-week modafinil treatment), checking UPDRS (and PSP scale as well if for PSP patient), stand-walk-sit, freezing of gait questionnaire, MoCA, anxiety scale and Epworth sleep scale at each visit before and 1 hour after the dopaminergic medication(s) (if the patient is on dopaminergic medication). Daily falls, freezing of gait and quality of life (by PDQ-39) over the past week prior to the clinical visit will also be checked.

A paired t-test will be used to compare the changes under each regimen with that at baseline, with primary outcome on gait difficulty of FOG frequency and severity, and secondary outcome on anxiety, cognition, UPDRS-III (plus PSP scale for PSP patients), and Epworth sleep scale (for modafinil trial) at dopaminergic medication off (after staying off the dopaminergic medication for over night) and on (1 hour after taking dopaminergic medication) state and quality of life assessment. The investigators want to see if the medications of different working mechanism, along or in combination, could improve the FOG and other motor symptoms, through the improvement of anxiety, cognitive dysfunction and wakening state at dopaminergic medications (for parkinsonism) off state and on state.

ELIGIBILITY:
Inclusion Criteria:

* Parkinsonian patient with Parkinson's disease per UK brain bank criteria 15,
* or PSP per SPSP-NINDS criteria 16,
* FOG at off or on dopaminergic medication or both.

Exclusion Criteria:

* Patients with psychosis,
* unable to walk without assistance,
* seizures,
* or allergy to any of these three medications on trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Freezing of Gait | From baseline to completion of drug regimen (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Changes in score of the stand-walk-sit test, compared to the baseline, at on and off PD medications status.
Freezing of Gait | From baseline to completion of drug regimen (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Changes in the score of the FOG questionnaire compared to the baseline, at on and off PD medications status.

SECONDARY OUTCOMES:
Change in anxiety | From baseline to completion of drug regiment (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Change in anxiety as measured by GDA-7 score compared to the baseline, at on and off PD medications status.
Change in cognition | From baseline to completion of drug regiment (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Change in cognition as measured by MoCA score compared to the baseline, at on and off PD medications status.
Change in symptom score/severity | From baseline to completion of drug regiment (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Change in symptom as measured by UPDRS or PSPRS score compared to the baseline, at on and off PD medications status.
Change in sleep quality | From baseline to completion of drug regiment (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Change in reported sleep quality as measured by the Epworth score compared to the baseline, at on and off PD medications status.
Change in quality of life | From baseline to completion of drug regiment (4 weeks of duloxetine, 2 weeks of duloxetine & donepezil, 2 weeks & 3 days modafinil)
  Change in reported quality of life as measured by QoL - PDQ-39 compared to the baseline, at on and off PD medications status.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Nutt JG, Bloem BR, Giladi N, Hallett M, Horak FB, Nieuwboer A. Freezing of gait: moving forward on a mysterious clinical phenomenon. Lancet Neurol. 2011 Aug;10(8):734-44. doi: 10.1016/S1474-4422(11)70143-0. PMID 21777828
- [Background] Shine JM, Matar E, Ward PB, Frank MJ, Moustafa AA, Pearson M, Naismith SL, Lewis SJ. Freezing of gait in Parkinson's disease is associated with functional decoupling between the cognitive control network and the basal ganglia. Brain. 2013 Dec;136(Pt 12):3671-81. doi: 10.1093/brain/awt272. Epub 2013 Oct 18. PMID 24142148
- [Background] Fasano A, Herman T, Tessitore A, Strafella AP, Bohnen NI. Neuroimaging of Freezing of Gait. J Parkinsons Dis. 2015;5(2):241-54. doi: 10.3233/JPD-150536. PMID 25757831
- [Background] Bohnen NI, Frey KA, Studenski S, Kotagal V, Koeppe RA, Scott PJ, Albin RL, Muller ML. Gait speed in Parkinson disease correlates with cholinergic degeneration. Neurology. 2013 Oct 29;81(18):1611-6. doi: 10.1212/WNL.0b013e3182a9f558. Epub 2013 Sep 27. PMID 24078735
- [Background] Lewitt PA. Norepinephrine: the next therapeutics frontier for Parkinson's disease. Transl Neurodegener. 2012 Jan 13;1(1):4. doi: 10.1186/2047-9158-1-4. PMID 23211006
- [Background] Pagano G, Rengo G, Pasqualetti G, Femminella GD, Monzani F, Ferrara N, Tagliati M. Cholinesterase inhibitors for Parkinson's disease: a systematic review and meta-analysis. J Neurol Neurosurg Psychiatry. 2015 Jul;86(7):767-73. doi: 10.1136/jnnp-2014-308764. Epub 2014 Sep 15. PMID 25224676
- [Background] Morgante F, Fasano A. Improvement with duloxetine in primary progressive freezing gait. Neurology. 2010 Dec 7;75(23):2130-2. doi: 10.1212/WNL.0b013e318200d7a3. No abstract available. PMID 21135389
- [Background] Nandi D, Jenkinson N, Stein J, Aziz T. The pedunculopontine nucleus in Parkinson's disease: primate studies. Br J Neurosurg. 2008;22 Suppl 1:S4-8. doi: 10.1080/02688690802448350. PMID 19085345
- [Background] Xie T, Vigil J, MacCracken E, Gasparaitis A, Young J, Kang W, Bernard J, Warnke P, Kang UJ. Low-frequency stimulation of STN-DBS reduces aspiration and freezing of gait in patients with PD. Neurology. 2015 Jan 27;84(4):415-20. doi: 10.1212/WNL.0000000000001184. Epub 2014 Dec 24. PMID 25540305
- [Background] Plaha P, Gill SS. Bilateral deep brain stimulation of the pedunculopontine nucleus for Parkinson's disease. Neuroreport. 2005 Nov 28;16(17):1883-7. doi: 10.1097/01.wnr.0000187637.20771.a0. PMID 16272872
- [Background] Mazzone P, Lozano A, Stanzione P, Galati S, Scarnati E, Peppe A, Stefani A. Implantation of human pedunculopontine nucleus: a safe and clinically relevant target in Parkinson's disease. Neuroreport. 2005 Nov 28;16(17):1877-81. doi: 10.1097/01.wnr.0000187629.38010.12. PMID 16272871
- [Background] Acar F, Acar G, Bir LS, Gedik B, Oguzhanoglu A. Deep brain stimulation of the pedunculopontine nucleus in a patient with freezing of gait. Stereotact Funct Neurosurg. 2011;89(4):214-9. doi: 10.1159/000326617. Epub 2011 May 20. PMID 21597312
- [Background] Garcia-Rill E, Kezunovic N, Hyde J, Simon C, Beck P, Urbano FJ. Coherence and frequency in the reticular activating system (RAS). Sleep Med Rev. 2013 Jun;17(3):227-38. doi: 10.1016/j.smrv.2012.06.002. Epub 2012 Oct 6. PMID 23044219